CLINICAL TRIAL: NCT02305680
Title: EPICOR Asia-China Extension. Long-term Follow-up of antithrombotIc Management Patterns in Acute Coronary Syndrome Patients in Asia-China Extension
Brief Title: Long-term Follow-up of antithrombotIc Management Patterns in Acute Coronary Syndrome Patients in Asia-China Extension
Acronym: EPICOR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00049; NIS-CCN-XXX-2014/1 (Other: Astrazeneca interal study number)
Record Dates: First submitted 2014-11-18; First posted 2014-12-03 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is to describe the long-term antithrombotic management patterns in a real-life setting for patients hospitalized with an acute coronary syndrome in China.

DETAILED DESCRIPTION:
This study is to describe the long-term (3 to 5 years after the acute coronary syndrome index event) antithrombotic management patterns in a real-life setting for patients hospitalized with an acute coronary syndrome (i.e. ST-segment Elevation Myocardial Infarction, Non-ST-segment Elevation Myocardial Infarction, Unstable Angina) in China.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been provided.
2. Contact Order Form has been provided
3. Aged 18 years or older.
4. Enrolled in EPICOR Asia study and completed the 2 year follow-up.

Exclusion Criteria:

1. Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language, psychiatric disturbances, alcohol or drug abuse).
2. Already included in the EPICOR Asia-China Extension observational study.
3. Presence of serious/severe co-morbidities in the opinion of the investigator which may limit short term (i.e. 6 month) life expectancy.
4. Current participation in an interventional clinical trial.
5. Patients receiving ticagrelor beyond 12 months and other off label use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a history of acute coronary syndromes in China
Sampling Method: Probability Sample
Enrollment: 2334 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Long-term antithrombotic management patterns in a real-life setting by assessing the medication and treatment prescribed by physicians | From 2 years after the acute coronary syndrome index event, assessed up to 5 years

SECONDARY OUTCOMES:
Clinical outcomes by record the number and type of cardiovascular and non-cardiovascular events | From 2 years after the acute coronary syndrome index event, assessed up to 5 years
Health care resource consumption and related costs by assessing the detail hospitalization and outpatient cost. | From 2 years after the acute coronary syndrome index event, assessed up to 5 years
Quality of life by assessing EQ-5D questionnaire. | 2 years,2.5years,3years,3.5years,4years,4.5years,5years after the acute coronary syndrome index event

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, Doctor, Principal Investigator — Peking University First Hospital
Locations (33):
- China (33):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Changzhi
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haerbin
  - Research Site, Hangzhou
  - Research Site, Hebei
  - Research Site, Jilin
  - Research Site, Jinan
  - Research Site, Jinzhong
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shihezi
  - Research Site, Taiyuan
  - Research Site, Tangshan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xining
  - Research Site, Xuzhou
  - Research Site, Yinchuan
  - Research Site, Yulin
  - Research Site, Zhengzhou
  - Research Site, Zhenjiang

REFERENCES:
- See also: D1843R00049 EPICOR CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3681&filename=D1843R00049_EPICOR_CSR%20Synopsis.PDF